CLINICAL TRIAL: NCT06288581
Title: Evaluating the Effectiveness of a U-shaped Toothbrush in Removing Plaque In Pre-school Children
Brief Title: U Shaped Toothbrush in Removing Plaque in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Damascus University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: UDDS-Pedo-02-2024
Record Dates: First submitted 2024-02-25; First posted 2024-03-01 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Dental Plaque
Keywords: U shaped toothbrush; Traditional toothbrush; Plaque removal; Oral hygiene; Pre-schooled children
MeSH Terms: conditions — Dental Plaque

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Traditional toothbrush group (Experimental): Children in this group will use a traditional brush first to clean their teeth then will use U shaped brush later.
  Interventions: Other: Traditional toothbrush group
- U shaped toothbrush group (Experimental): children in this group will use a U-shaped brush first to clean their teeth then will use traditional brush later
  Interventions: Other: U shaped toothbrush group

INTERVENTIONS:
Other: Traditional toothbrush group — Children in this group will use a traditional brush with a traditional toothpaste first to clean their teeth then after 30 days they will use a U shaped brush with a traditional toothpaste for another 30 days.
  Arms: Traditional toothbrush group
Other: U shaped toothbrush group — Children in this group will use a U shaped brush with a traditional toothpaste first to clean their teeth then after 30 days they will use a traditional brush with a traditional toothpaste for another 30 days.
  Arms: U shaped toothbrush group

SUMMARY:
The aim of this study is to evaluate the effectiveness of a U-shaped toothbrush in removing plaque in preschool children which can be a simple, acceptable, and effective way to remove plaque in children in order to improve their oral health in the absence of parental supervision.

Children accepted in the study will be randomly divided into two groups:

The traditional toothbrush group and the U-shaped toothbrush group, All children aged four to five years will have their plaque assessed with the Turesky Modified Quigley Hein Index (TMQH)

DETAILED DESCRIPTION:
This study will evaluate the effectiveness U-shaped toothbrush in removing plaque and improving oral health. Children were randomly assigned to one of the following groups:

Group A: children in this group will use a traditional brush first to clean their teeth then will use U shaped brush later.

Group B: children in this group will use a U-shaped brush first to clean their teeth then will use a traditional brush later The plaque will be assessed by a blinded evaluator using the Turesky Modified Quigley Hein index (TMQH) in both groups at 4 different times(T0): before brush (T1): after brush (T2): a week after use (T3): a month of use The toothbrush will be changed after one month of use.

ELIGIBILITY:
Inclusion Criteria:

Medically free children. Complete temporary occlusion (no missing temporary teeth). The parents' approval for the child to enter the study.

Exclusion Criteria:

Children with limited ability to communicate. Children with motor disabilities.

Ages: 4 Years to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2024-02-01 (Actual); Primary Completion 2024-05-01 (Actual); Study Completion 2024-08-15 (Actual)

PRIMARY OUTCOMES:
Changing in plaque index | Plaque index will be measured before brushing (T0) and after brushing in both groups on the first day (T1), a week after use (T2), and after a month of use (T3) with each toothbrush
  0 No plaque,1 Isolated flecks of plaque at the gingival margin, 2 A continuous band of plaque up to 1mm at the gingival margin, 3 Plaque greater than 1mm in width and covering up to one third of the tooth surface, 4 Plaque covering from one thirds to two thirds of the tooth surface, and 5 Plaque covering more than two thirds of the tooth surface

CONTACTS AND LOCATIONS:
Locations (1):
- Damascus University, Damascus, Syria

IPD SHARING:
Plan to Share IPD: No
only with contacting the main researcher